CLINICAL TRIAL: NCT02323191
Title: Open-Label, Multicenter, Dose Escalation Phase Ib Study With Expansion Phase to Evaluate the Safety, Pharmacokinetics, and Activity of RO5509554 (Emactuzumab) and MPDL3280A (Atezolizumab) Administered in Combination in Patients With Advanced Solid Tumors
Brief Title: A Study of Emactuzumab and Atezolizumab Administered in Combination in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP29428; 2014-002428-29 (EudraCT Number); RG7155 (Other: Roche)
Record Dates: First submitted 2014-12-05; First posted 2014-12-23 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Solid Cancers
MeSH Terms: interventions — atezolizumab; emactuzumab

ARMS (2):
- Part 1 (Dose-finding): Emactuzumab + Atezolizumab (Experimental): Participants will receive escalating doses of emactuzumab along with atezolizumab every 3 weeks (q3w).
  Interventions: Drug: Atezolizumab; Drug: Emactuzumab
- Part 2 (Expansion): Emactuzumab + Atezolizumab (Experimental): Participants will receive emactuzumab at or below the MTDs for the combination treatments that are determined during Part 1 along with atezolizumab.
  Interventions: Drug: Atezolizumab; Drug: Emactuzumab

INTERVENTIONS:
Drug: Atezolizumab — Participants will receive atezolizumab intravenously at a fixed dose of 1200 milligram (mg) q3w.
  Other Names: MPDL3280A, TECENTRIQ
Drug: Emactuzumab — Participants will receive emactuzumab intravenously in ascending dose levels with a starting dose of 500 mg.
  Other Names: RO5509554

SUMMARY:
This Phase 1, open-label, multicenter, global study will evaluate the safety, pharmacokinetics, and activity of emactuzumab and atezolizumab administered in combination in participants with selected locally advanced or metastatic solid tumors that are not amenable to standard treatment.

Participants who receive emactuzumab and atezolizumab will continue to receive study drug as long as they experience clinical benefit in the opinion of the investigator or until unacceptable toxicity or symptomatic deterioration attributed to disease progression as determined by the investigator after an integrated assessment of radiographic data, biopsy results (if available), and clinical status, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status 0 or 1
* Participants must have histologically confirmed diagnosis of locally advanced and/or metastatic triple negative breast cancer, ovarian cancer, bladder cancer, gastric cancer, or soft tissue sarcoma, with exceptions defined in the exclusion criteria
* Measurable disease at baseline as per RECIST version 1.1
* Life expectancy of greater than or equal to (>=) 16 weeks
* Adequate bone marrow, liver, cardiac, and renal function
* Negative serum pregnancy test within 7 days prior to study treatment in premenopausal women and women less than or equal to (<=) 12 months post-menopause. Postmenopausal state is defined as amenorrhea for greater than (>) 12 months.

Exclusion Criteria:

* Allergy or hypersensitivity to components of the emactuzumab formulation or to components of the atezolizumab formulation
* Active or untreated central nervous system (CNS) metastases as determined by computed tomography (CT) or magnetic resonance imaging evaluation during screening (within 28 days before C1D1) and prior radiographic assessments. Participants with radiographically stable, asymptomatic previously irradiated lesions are eligible provided participant is >= 4 weeks beyond completion of cranial irradiation and >= 3 weeks off of corticosteroid therapy. Participants with metastases to the brain stem, midbrain, pons, medulla, or within 10 millimeter (mm) of the optic apparatus (optic nerves and chiasm) are completely excluded
* Leptomeningeal disease
* History of or active autoimmune disease
* Evidence of significant, uncontrolled concomitant diseases, which could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina) or pulmonary disease (including obstructive pulmonary disease and history of symptomatic bronchospasm)
* Any approved anti-cancer therapy, including chemotherapy or hormonal therapy, within 3 weeks prior to initiation of study treatment, with the exceptions provided in the protocol
* Prior corticosteroids as anti-cancer therapy within a minimum of 14 days of first receipt of study drug
* Prior toxicities from chemotherapy, radiotherapy, and other anti-cancer therapies, including immunotherapy that have not regressed to Grade <=1 severity (Common Terminology Criteria for Adverse Events [CTCAE] v4.03, or later versions)
* History of human immunodeficiency virus (HIV)
* Participants with active hepatitis B, active hepatitis C, or active tuberculosis
* Participant has had pulmonary embolism or any other thrombo-embolic event within 6 months prior to study entry
* Participants has a history of hematological malignancy within the last 5 years prior to study entry
* Treatment with systemic immunosuppressive medications - Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2015-01-19 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose Limiting Toxicities (DLTs) | 21 days
Maximum Tolerated Dose (MTD) of Emactuzumab | 21 days
Percentage of Participants With Adverse Events (AEs) | Baseline up to 3 years

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Emactuzumab | predose (-4 h) on Day 1 of Cycle 1 up to approximately 3 years (detailed timeframe provided in measure description)
  predose (-4 hours [h]) and 0.5h post end of infusion (90 minutes infusion) on Days (D) 1 of Cycle (C) 1, 2, 3, 4, 5, 6, all subsequent cycles (Cycle Length=21 days) until disease progression (up to approximately 3 years); 5h postdose on D1 of C1; postdose on D2, D4 or D5, D8, D15 of C1, C2, C4; D12, D19 of C1, C4; 44 and 120 days post last infusion; 28 day follow-up visit (up to approximately 3 years)
Maximum Observed Plasma Concentration (Cmax) of Atezolizumab | predose (-4 h) on D1 of C1, C2, C3, C4, C6, then every 8 cycles (Cycle Length=21 days); 0.5h post end of infusion (60 minutes infusion) on D1 of C1; 120 days post last infusion (up to approximately 3 years)
Minimum Observed Plasma Trough Concentration (Cmin) of Emactuzumab | predose (-4 h) on D1 of C2, C3, C4, C5, C6, all subsequent cycles (Cycle Length=21 days) until disease progression (up to approximately 3 years)
Minimum Observed Plasma Trough Concentration (Cmin) of Atezolizumab | predose (-4 h) on D1 of C1, C2, C3, C4, C6, then every 8 cycles (Cycle Length=21 days)
Area under the Concentration-Time Curve (AUC) of Emactuzumab | predose (-4 h) on Day 1 of Cycle 1 up to approximately 3 years (detailed timeframe provided in measure description)
  predose (-4 h) and 0.5h post end of infusion (90 minutes infusion) on D1 of C1, C2, C3, C4, C5, C6, all subsequent cycles (Cycle Length=21 days) until disease progression (up to approximately 3 years); 5h postdose on D1 of C1; postdose on D2, D4 or D5, D8, D15 of C1, C2, C4; D12, D19 of C1, C4; 44 and 120 days post last infusion; 28 day follow-up visit (up to approximately 3 years)
Total Clearance (CL) of Emactuzumab | predose (-4 h) and 0.5h post end of infusion (90 minutes infusion) on D1 of C1, C4 (Cycle Length=21 days); 5h postdose on D1 of C1; postdose on D2, D4 or D5, D8, D12, D15, D19 of C1, C4
Volume of Distribution at Steady State (Vss) of Emactuzumab | predose (-4 h) and 0.5h post end of infusion (90 minutes infusion) on D1 of C1, C4 (Cycle Length=21 days); 5h postdose on D1 of C1; postdose on D2, D4 or D5, D8, D12, D15, D19 of C1, C4
Accumulation Ratio (Rac) of Emactuzumab | predose (-4 h) and 0.5h post end of infusion (90 minutes infusion) on D1 of C1, C4 (Cycle Length=21 days); 5h postdose on D1 of C1; postdose on D2, D4 or D5, D8, D12, D15, D19 of C1, C4
Terminal Elimination Half-life (t1/2) of Emactuzumab | predose (-4 h) and 0.5h post end of infusion (90 minutes infusion) on D1 of C1, C4 (Cycle Length=21 days); 5h postdose on D1 of C1; postdose on D2, D4 or D5, D8, D12, D15, D19 of C1, C4
Emactuzumab Concentration at the time of Tumor Progression (Cprog) | predose (-4 h) on Day 1 of Cycle 1 up to approximately 3 years (detailed timeframe provided in measure description)
  predose (-4 h) and 0.5h post end of infusion (90 minutes infusion) on D1 of C1, C2, C3, C4, C5, C6, all subsequent cycles (Cycle Length=21 days) until disease progression (up to approximately 3 years); 5h postdose on D1 of C1; postdose on D2, D4 or D5, D8, D15 of C1, C2, C4; D12, D19 of C1, C4; 44 and 120 days post last infusion; 28 day follow-up visit (up to approximately 3 years)
Emactuzumab Concentration at the Time of Tumor Response (Complete Response/Partial Response) | predose (-4 h) on Day 1 of Cycle 1 up to approximately 3 years (detailed timeframe provided in measure description)
  predose (-4 h) and 0.5h post end of infusion (90 minutes infusion) on D1 of C1, C2, C3, C4, C5, C6, all subsequent cycles (Cycle Length=21 days) until disease progression (up to approximately 3 years); 5h postdose on D1 of C1; postdose on D2, D4 or D5, D8, D15 of C1, C2, C4; D12, D19 of C1, C4; 44 and 120 days post last infusion; 28 day follow-up visit (up to approximately 3 years)
Emactuzumab Concentration at the Time of Infusion-related Reaction (IRR) or Hypersensitivity Reaction | predose (-4 h) on Day 1 of Cycle 1 up to approximately 3 years (detailed timeframe provided in measure description)
  predose (-4 h) and 0.5h post end of infusion (90 minutes infusion) on D1 of C1, C2, C3, C4, C5, C6, all subsequent cycles (Cycle Length=21 days) until disease progression (up to approximately 3 years); 5h postdose on D1 of C1; postdose on D2, D4 or D5, D8, D15 of C1, C2, C4; D12, D19 of C1, C4; 44 and 120 days post last infusion; 28 day follow-up visit (up to approximately 3 years)
Change From Baseline in Tumor-Associated Macrophages (TAMs) Levels in Paired-Tumor Biopsies at Specified Timepoints | Baseline (predose [-4 h] on D1 of C2; Cycle Length=21 days), at disease progression (up to approximately 3 years)
Change From Baseline in Dermal Macrophages Levels in Paired Skin Biopsies at Specified Timepoints | Baseline, D15 of C1 (Cycle Length=21 days)
Change From Baseline in Circulating Cluster of Differentiation (CD) 14DimCD16high Monocytes Levels in Peripheral Blood at Specified Timepoints | Baseline up to approximately 3 years (detailed timeframe provided in measure description)
  Baseline (predose [-4 h] on D1 of C1), predose [-4 h] on D1 of C2, C3, C5, then every other cycle (Cycle Length=21 days) until disease progression (up to approximately 3 years); postdose on D2, D8, D15 of C1, C2; D4 or D5 of C1; 44 days post last infusion (up to approximately 3 years)
Percentage of Participants With Anti-therapeutic Antibodies to Emactuzumab | predose (-4 h) on D1 of C1, C2, C3, C4, C6, all subsequent cycles (Cycle Length=21 days) until disease progression (up to approximately 3 years), 44 and 120 days post last infusion, 28 day follow-up visit (up to approximately 3 years)
Percentage of Participants With Anti-therapeutic Antibodies to Atezolizumab | predose (-4 h) on D1 of C1, C2, C3, C4, C6, then every 8 cycles (Cycle Length=21 days; up to approximately 3 years), 120 days post last infusion (up to approximately 3 years)
Percentage of Participants With Best Overall Response as Determined Using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Baseline up to disease progression or death, whichever occurs first (assessed up to approximately 3 years)
Percentage of Participants With Best Overall Response as Determined Using Modified RECIST | Baseline up to disease progression or death, whichever occurs first (assessed up to approximately 3 years)
Percentage of Participants With Objective Response as Determined Using RECIST v1.1 | Baseline up to disease progression or death, whichever occurs first (assessed up to approximately 3 years)
Percentage of Participants With Objective Response as Determined Using Modified RECIST | Baseline up to disease progression or death, whichever occurs first (assessed up to approximately 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- United States (5):
  - Yale Cancer Center; Medical Oncology, New Haven, Connecticut
  - Massachusetts General Hospital., Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber - Harvard, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center Breast & Imaging Center, New York, New York
- Cliniques Universitaires St-Luc, Brussels, Belgium
- France (3):
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif
- Spain (3):
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Centro Integral Oncológico Clara Campal Ensayos Clínicos START, Madrid

REFERENCES:
- [Derived] Gomez-Roca C, Cassier P, Zamarin D, Machiels JP, Perez Gracia JL, Stephen Hodi F, Taus A, Martinez Garcia M, Boni V, Eder JP, Hafez N, Sullivan R, Mcdermott D, Champiat S, Aspeslagh S, Terret C, Jegg AM, Jacob W, Cannarile MA, Ries C, Korski K, Michielin F, Christen R, Babitzki G, Watson C, Meneses-Lorente G, Weisser M, Ruttinger D, Delord JP, Marabelle A. Anti-CSF-1R emactuzumab in combination with anti-PD-L1 atezolizumab in advanced solid tumor patients naive or experienced for immune checkpoint blockade. J Immunother Cancer. 2022 May;10(5):e004076. doi: 10.1136/jitc-2021-004076. PMID 35577503